CLINICAL TRIAL: NCT04848558
Title: A Phase 1 Double-Blind, Placebo-Controlled, Single- and Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneous Nipocalimab in Healthy Male and Female Participants
Brief Title: A Study of Nipocalimab in Healthy Male and Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CR108993; 2020-005892-10 (EudraCT Number); 80202135EDI1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Single Dose Cohorts (Experimental): Participants will receive subcutaneous (SC) injection or intravenous (IV) infusion of nipocalimab or placebo in single ascending doses on Day 1 in Cohorts 1-6 and SC administration in optional Cohorts 7-8.
  Interventions: Drug: Nipocalimab; Other: Placebo
- Part 2: Multiple Dose Cohorts (Experimental): Participants will receive up to 4 weekly SC injections of nipocalimab or placebo on Days 1, 8, 15, and 22 in Cohort 1 or 4 biweekly SC injections on Days 1, 15, 29, and 43 in optional Cohort 2.
  Interventions: Drug: Nipocalimab; Other: Placebo

INTERVENTIONS:
Drug: Nipocalimab — Participants will receive IV infusion or SC injection of nipocalimab.
  Other Names: JNJ-80202135
Other: Placebo — Participants will receive IV infusion or SC injection of placebo.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single and multiple doses of nipocalimab following subcutaneous (SC) administration compared with intravenous (IV) administration in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening
* Healthy on the basis of clinical laboratory tests performed at screening
* Continuous non-smoker
* A woman of childbearing potential must have a negative pregnancy test
* It is recommended that participants are up to date on all age appropriate vaccinations prior to screening as per routine local medical guidelines

Exclusion Criteria:

* Has a history of liver or renal insufficiency; cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Currently has a malignancy or has a history of malignancy within 3 years before screening
* Known allergies, hypersensitivity, or intolerance to nipocalimab or its excipients
* Has received a live vaccine within 3 months prior to screening or has a known need to receive a live vaccine during the study, or within at least 3 months after the last administration of study intervention in this study
* Shows evidence of an active or chronic hepatitis B infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to Day 85
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Percentage of Participants with Serious Adverse Event (SAE) | Up to Day 85
  A SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.
Percentage of Participants with Reasonably Related AEs | Up to Day 85
  Percentage of participants with reasonably related AEs will be reported. Reasonably related AE is an AE that has a casual relationship with the pharmaceutical/biological agent under study.
Percentage of Participants with AEs Leading to Discontinuation of Study Intervention | Up to Day 85
  Percentage of participants with AEs leading to discontinuation of study intervention will be reported. The participants were discontinued from the study by the investigator if the safety reasons or tolerability reasons such as an AE, it is in the best interest of the participant to discontinue study intervention.
Percentage of Participants with Adverse Events of Special Interest (AESIs) | Up to Day 85
  Percentage of participants with AESIs will be reported. Treatment-emergent AEs associated with the following situations are considered as AESI; a) severe or medically significant or immediately life-threatening infections requiring intravenous (IV) anti-infective or operative/invasive intervention or requiring hospitalization or prolongation of existing hospitalization; b) hypoalbuminemia with albumin less than (<) 20 grams per liter (g/L). Treatment-emergent AEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Number of Participants with Vital Signs Abnormalities | Up to Day 85
  Number of participants with vital signs abnormalities including body temperature, pulse/heart rate, respiratory rate, blood pressure will be reported.
Number of Participants with Electrocardiogram (ECG) Abnormalities | Up to Day 85
  Number of participants with ECG abnormalities will be reported.
Number of Participants with Clinical Laboratory Abnormalities | Up to Day 85
  Number of participants with clinical laboratory abnormalities related to hematology, serum chemistry and urinalysis will be reported.
Number of Participants with Subcutaneous (SC) Injection-site Reactions | Up to Day 85
  Number of participants with SC injection-site reactions will be reported. An injection-site reaction is any AE at a SC study intervention injection-site.

SECONDARY OUTCOMES:
Serum Concentration of Nipocalimab | Up to Day 85
  Serum samples will be analyzed to determine concentrations of nipocalimab using a validated, specific, and sensitive immunoassay method.
Change from Baseline in Immunoglobulin (Ig) Levels Over Time | Baseline to Day 85
  Change from baseline in Ig levels over time will be reported.
Number of Participants with Antibodies to Nipocalimab | Up to Day 85
  Number of participants with anti-drug antibodies to nipocalimab will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinicaltrials/ transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency